CLINICAL TRIAL: NCT05712655
Title: Electromyographic Activity of Masticatory Muscles in Post-pubertal Females With Forward Head Posture and Temporomandibular Disorders: An Observational Trial
Brief Title: Masticatory Muscles Electromyography in Post-pubertal Females With Forward Head Posture and Temporomandibular Disorders
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa A. Osman, Assistant Professor, Cairo University
Other Study IDs: P.T.REC/012/002660
Record Dates: First submitted 2023-01-22; First posted 2023-02-03 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Head Pain; TMJ Disorder
Keywords: Forward head posture; Temporomandibular disorders; Masticatory muscles; Electromyography; post-pubertal females
MeSH Terms: conditions — Headache; Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Post-pubertal females with forward head posture and temporomandibular disorders
  Interventions: Other: Measurement of bilateral electromyographic activity of Masseter and Anterior Temporalis muscles.
- Control group: Post-pubertal females with neutral head posture and with no temporomandibular disorders
  Interventions: Other: Measurement of bilateral electromyographic activity of Masseter and Anterior Temporalis muscles.

INTERVENTIONS:
Other: Measurement of bilateral electromyographic activity of Masseter and Anterior Temporalis muscles. — Assessment was done by surface electromyography (sEMG) device.

SUMMARY:
The aim of this study was to evaluate masticatory muscle electrical activity in post-pubertal females with forward head posture (FHP) and temporomandibular disorders (TMD) as well as in post-pubertal females with neutral head posture and with no temporomandibular disorders.

DETAILED DESCRIPTION:
It has been demonstrated by a previous study that a strong relationship exists between forward head posture and temporomandibular disorders and that individuals with forward head posture and temporomandibular disorders exhibit alterations in masticatory muscle electromyographic activity either as a result of the disorder itself or due to a compensatory mechanism associated with the symptoms of temporomandibular disorders . As a consequence, the aim of the study was to evaluate the electromyographic activity of the masticatory muscles in post-pubertal females with forward head posture and temporomandibular disorders as well as in post-pubertal females with neutral head posture and with no temporomandibular disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age ranging from 17 to 22 years.
* Body mass index ranging from 18 to 25 kg/m2.
* Having a normal menstrual cycle.
* Spending four to six hours per day with bad posture on computer, laptop or smart phones.
* Fully dentate subjects.

Exclusion Criteria:

* Having dental loss, acquired dental anomalies, current use of dental prostheses, malocclusion, sleep bruxism.
* Having inflammatory diseases of the face or jaw, fibromyalgia, or any fractures or surgeries in the orofacial or neck areas.

Ages: 17 Years to 22 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes
Study Population: They were invited to participate in the study through flyers and social media invitations
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Electromyographic (EMG) activity of masticatory muscles | 8 months
  Measurement of bilateral EMG activity of Masseter and Anterior Temporalis muscles

SECONDARY OUTCOMES:
Measurement of cranivertebral angle (CVA) | 8 months
  Photographic assessment of cranivertebral angle.
Assessment of research Diagnostic criteria for temporomandibular Disorders (RDC/TMDS) | 8 months
  Temporomandibular disorders were assessed through the research Diagnostic criteria for temporomandibular Disorders (RDC/TMDS).

CONTACTS AND LOCATIONS:
Overall Officials: Amel M Yousef, Professor, Principal Investigator — Physical Therapy for Woman's Health, Faculty of physical therapy, Cairo University, Giza, Egypt.
Locations (1):
- Nasser Institute for research and treatment, Cairo, Egypt